CLINICAL TRIAL: NCT00081107
Title: A Phase II Study of KOS-862, Administered Intravenously Weekly for 3 Weeks Every 4 Weeks, in Patients With Non-Small Cell Lung Cancer Who Have Progressed Following Initial Therapy for Advanced or Metastatic Disease
Brief Title: Epothilone D in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer That Has Not Responded to Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 03-134; CDR0000358910 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-N017352; KOS-201
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — desoxyepothilone B

INTERVENTIONS:
Drug: epothilone D

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epothilone D, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well epothilone D works in treating patients with stage IIIB or stage IV non-small cell lung cancer that has not responded to platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of epothilone D, in terms of confirmed objective response rate, in patients with stage IIIB or IV non-small cell lung cancer who failed prior initial platinum-containing chemotherapy.

Secondary

* Determine the safety of this drug in these patients.
* Determine the response duration in patients who achieve complete response or partial response, time to tumor progression, and survival in patients treated with this drug.
* Compare the power associated with the estimated treatment effect of this drug in these patients vs standard treatment.
* Correlate efficacy and safety with plasma concentrations of this drug and its major metabolites in these patients.

OUTLINE: This is a multicenter, open-label study.

Patients receive epothilone D IV over 90 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 33-85 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB* or IV disease NOTE: *Due to malignant pleural effusion or supraclavicular lymph node involvement only
* Previously treated with maximally feasible surgical resection and/or radiotherapy for initial disease
* Failed 1 prior platinum-containing chemotherapy regimen for advanced or metastatic disease due to disease progression or treatment toxicity
* At least 1 site of unidimensionally measurable disease by physical exam or radiography
* No known CNS metastases or leptomeningeal metastases requiring corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 75,000/mm^3

Hepatic

* AST ≤ 2.5 times upper limit of normal (ULN) (5 times ULN for patients with hepatic metastases)
* Alkaline phosphatase ≤ 5 times ULN
* Bilirubin ≤ 1.8 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No personal or family history of congenital long QT syndrome
* No QTc interval > 450 msec (males) or > 470 msec (females) by ECG

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No preexisting neuropathy ≥ grade 2
* No other malignancy within the past 5 years except for the following:

  * Cured basal cell skin cancer
  * Carcinoma in situ of the cervix or urinary bladder
  * Stage T1 or T2 prostate cancer with prostate-specific antigen < 2 ng/mL
* No hypersensitivity reaction ≥ grade 3 to prior Cremophor-containing therapy
* No infection requiring parenteral or oral anti-infective therapy
* No weight loss of ≥ 10% within the past 3 months
* No altered mental status or psychiatric illness that would preclude giving informed consent
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent granulocyte-macrophage colony-stimulating factor (sargramostim [GM-CSF])
* No concurrent routine prophylactic granulocyte colony-stimulating factor (filgrastim [G-CSF])

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* At least 3 weeks since prior surgery and recovered

Other

* Prior adjuvant or neoadjuvant therapy allowed
* Prior radiosensitizers allowed
* At least 2 weeks since prior gefitinib
* More than 3 weeks since prior investigational agents (therapeutic or diagnostic)
* No other concurrent investigational agents
* No other concurrent anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States